CLINICAL TRIAL: NCT02211521
Title: Randomized, Double Blind, Comparison Clinical Trial to Test the Efficacy and Safety of Intraarticular Injection of Autologous Platelet-rich Plasma (PRP) for the Treatment of Osteoarthritis of the Knee Joint
Brief Title: Comparison of Autologous Platelet-rich Plasma With Hyaluronic Acid for the Treatment of Osteoarthritis of the Knee Joint
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, ChulWon Ha, Professor of Department of Orthopaedic Surgery, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-12-056
Record Dates: First submitted 2014-07-18; First posted 2014-08-07 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, platelet-rich plasma, hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRP group (Experimental): Patients randomized to this group of treatment will receive 1 blinded knee intra-articular injections of autologous Platelet-Rich Plasma (3ml).
  Interventions: Biological: PRP
- Hyaloronan group (Active Comparator): Patients randomized to this group of treatment will receive 1 blinded knee intra-articular injections of hyaluronic acid (3ml)
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Biological: PRP — 3ml of PRP
  Other Names: GPS III, Biomet Biologics, Warsaw, Ind, USA
  Arms: PRP group
Drug: Hyaluronic acid — 3ml hyaluronic acid
  Other Names: LBSA0103, 60 mg/3ml, LG Life Sciences, Korea
  Arms: Hyaloronan group

SUMMARY:
The purpose of this study is to compare the efficacy of platelet-rich plasma versus hyaluronic acid intra-articular injections for the treatment of osteoarthritis of knee joint.

The hypothesis is that PRP intra-articular injection is comparable or even better than hyaluronic acid injection.

DETAILED DESCRIPTION:
Osteoarthritis (OA) has a significant impact on our society. The limited regenerative capacity of cartilage is part of this problem. Existing degenerative lesions lead to accelerated deterioration of the articular (joint) surface leading to end-stage arthritis. In particular, the most recent knowledge regarding tissue biology highlights a complex regulation of growth factors (GFs) for the normal tissue structure and the reaction to tissue damage. The influence of GFs on cartilage repair is now widely investigated in vitro and in vivo. Platelet Rich Plasma (PRP) is a simple, low- cost and minimally- invasive method that allows one to obtain a natural concentrate of autologous GFs from the blood, and it is increasingly applied in the clinical practice to treat knee degenerative pathology, such as chondropathy and early OA. The biological rational of PRP is that platelets contain storage pools of GFs, cytokines, chemokines and many other mediators.Although its widespread application, there are little high level studies in the literature to demonstrate the real efficacy of PRP.

The investigators hypothesized that intra-articular injections of PRP to treat knee osteoarthritis could determine pain relief and recovery of knee function with overall clinical outcome comparable or even better than viscosupplementation, which is a common injective approach applied in this kind of pathology. To this purpose the investigators designed a double blind randomized controlled trial comparing PRP vs viscosupplementation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis of knee (by American College of Rheumatology Criteria) and Kellgren-Lawrence grade I ~ III
* More than 40 out of 100-mm VAS scale for pain at screening and baseline
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Patients with Hb values < 10 g/dl and platelet values < 100,000/ul
* Patients with a current or medical history of autoimmune disease
* Recent fever ( within 2 weeks) or serious illness
* Local infection at the site of the procedure
* Corticosteroid injection at treatment site within 1 month
* Systematic use of corticosteroids within 2 weeks
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* Patients who have been administered with immunosuppressants within the past 6 weeks
* Patients who are enrolled in any other clinical trials within 4 weeks
* Patients who the principal investigator considers inappropriate for participation in the clinical trial for reasons other than those listed above

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in International Knee Documentation Committee subjective score at week 24 | Baseline, Week 24
  International Knee Documentation Committee subjective score for both groups

SECONDARY OUTCOMES:
Change from baseline in VAS (Visual Analogue scale) for pain during walking | Baseline, Week 6, Week 12, Week 24
  VAS (Visual Analogue scale) for pain during walking for both groups of treatment
Change from baseline in Western Ontario and McMaster Universities Arthritis Index | Baseline, Week 6, Week 12, Week 24
  Western Ontario and McMaster Universities Arthritis Index variation for both groups
  Subscale analysis of pain, stiffness, function also contain
Number of Participants with Adverse Events | Week 6, Week 12, Week 24
  All adverse events included
Change from baseline in Samsung Medical Center Patellofemoral score (SMC patellofemoral score) | Baseline, Week 6, Week 12, Week 24
  Samsung Medical Center Patellofemoral score for both groups of treatment
Patient global assessment | Week 6, Week 12, Week 24
  Patient global assessment was evaluated for improvement of symptoms using 100mm VAS.
Change from baseline in International Knee Documentation Committee subjective score at week 6, week 12 | Baseline, Week 6, Week 12
  International Knee Documentation Committee subjective score for both groups

OTHER OUTCOMES:
Level of white blood cell count of platelet rich plasma | baseline
  Assessment of level of WBC, platelet and several growth factors of platelet rich plasma Assessment of level of white blood cell count of platelet rich plasma
Level of platelet of platelet rich plasma | baseline
  Assessment of level of platelet of platelet rich plasma
Level of growth factors of platelet rich plasma | baseline
  Assessment of level several growth factors of platelet rich plasma (platelet derived growth factor, transforming growth factor -b1, vascular endothelial growth factor, epidermal growth factor, fibroblast growth factor etc)

CONTACTS AND LOCATIONS:
Overall Officials: Chul-WOn Ha, MD, PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Cerza F, Carni S, Carcangiu A, Di Vavo I, Schiavilla V, Pecora A, De Biasi G, Ciuffreda M. Comparison between hyaluronic acid and platelet-rich plasma, intra-articular infiltration in the treatment of gonarthrosis. Am J Sports Med. 2012 Dec;40(12):2822-7. doi: 10.1177/0363546512461902. Epub 2012 Oct 25. PMID 23104611
- [Background] Spakova T, Rosocha J, Lacko M, Harvanova D, Gharaibeh A. Treatment of knee joint osteoarthritis with autologous platelet-rich plasma in comparison with hyaluronic acid. Am J Phys Med Rehabil. 2012 May;91(5):411-7. doi: 10.1097/PHM.0b013e3182aab72. PMID 22513879
- [Background] Kon E, Mandelbaum B, Buda R, Filardo G, Delcogliano M, Timoncini A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma intra-articular injection versus hyaluronic acid viscosupplementation as treatments for cartilage pathology: from early degeneration to osteoarthritis. Arthroscopy. 2011 Nov;27(11):1490-501. doi: 10.1016/j.arthro.2011.05.011. Epub 2011 Aug 10. PMID 21831567
- [Background] Sundman EA, Cole BJ, Karas V, Della Valle C, Tetreault MW, Mohammed HO, Fortier LA. The anti-inflammatory and matrix restorative mechanisms of platelet-rich plasma in osteoarthritis. Am J Sports Med. 2014 Jan;42(1):35-41. doi: 10.1177/0363546513507766. Epub 2013 Nov 5. PMID 24192391
- [Derived] Park YB, Kim JH, Ha CW, Lee DH. Clinical Efficacy of Platelet-Rich Plasma Injection and Its Association With Growth Factors in the Treatment of Mild to Moderate Knee Osteoarthritis: A Randomized Double-Blind Controlled Clinical Trial As Compared With Hyaluronic Acid. Am J Sports Med. 2021 Feb;49(2):487-496. doi: 10.1177/0363546520986867. PMID 33523756